CLINICAL TRIAL: NCT04234542
Title: Is Low Level Laser Therapy (LLLT) Effective for Reducing Pain Experienced by Women With Provoked Vestibulodynia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: BioFlexTM Laser Therapy (Unknown)
Responsible Party: Principal Investigator, Dr. Linda McLean, Professor in the School of Rehabilitation Sciences at the University of Ottawa., University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-01-19-2367
Record Dates: First submitted 2020-01-09; First posted 2020-01-21 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Provoked Vestibulodynia
Keywords: vulvar pain; pelvic floor; low level laser therapy; laser; transcranial magnetic stimulation; electromyography
MeSH Terms: conditions — Vulvodynia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Level Laser Therapy Group (Experimental): 15 treatments will be provided over a 12 week period using a protocol developed in collaboration with BioFlexTM Laser. Each treatment will last approximately 45 minutes and will include the laser array first being applied to the skin overlying the sacral spine in a horizontal placement then in oblique placement bilaterally (red and infrared light) while a laser probe is applied over the base of the spine (red and infrared light). Next, the array will be applied to the surface of the perineum (red and infrared light) and the focal probe will be applied to painful sites on the perineum. Finally, the infrared light probe will be applied to the skin overlying branches of the pudendal nerve. All the stages will involve use of the same array and probe placement, but at each stage the dosage will be increased according to the BioFlex protocol. During teach treatment session, women will listen to an audio recording of a mindfulness-based meditation on CD through noise cancelling headphones.
  Interventions: Other: Low Level Laser Therapy
- Sham Low Level Laser Therapy Group (Sham Comparator): 15 treatments will be provided over a 12 week period using the same protocol developed in collaboration with BioFlexTM Laser, but at an intensity of 1% output for all sites and at all stages. Each treatment will last approximately 45 minutes. At each visit, the laser array will first be applied to the skin overlying the sacral spine in a horizontal then oblique placement bilaterally (red and infrared light) concurrently with a laser probe applied over the base of the spine (red and infrared light). Next, the array will be applied to the surface of the perineum (red and infrared light), followed by treatment at specific painful sites using the red light probe. Finally, the infrared light probe will be applied to the skin overlying branches of the pudendal nerve. Participants randomized to this group will listen to an audio recording of a mindfulness-based meditation on CD through noise cancelling headphones while receiving the sham laser treatment.
  Interventions: Other: Sham Low Level Laser Therapy

INTERVENTIONS:
Other: Low Level Laser Therapy — Each stage will follow this sequence of applications: (1) spine application (DUO-240 red and infrared array in a horizontal placement and 2 oblique placements bilaterally + LDR-100 laser probe + LDI-200 laser probe), (2) perineum application (DUO-240 red and infrared array in the surface of the perineum + LDR-100 probe) and (3) overlying branches of the pudendal nerve at the lateral perineum (LDI-200 probe). Parameters of frequency and duty cycle will be increased along with intensity as the stages progress.
  Other Names: photobiomodulation
  Arms: Low Level Laser Therapy Group
Other: Sham Low Level Laser Therapy — Each stage will follow this sequence of applications: (1) spine application (DUO-240 red and infrared array in a horizontal placement and 2 oblique placements bilaterally + LDR-100 laser probe + LDI-200 laser probe), (2) perineum application (DUO-240 red and infrared array in the surface of the perineum + LDR-100 probe) and (3) overlying branches of the pudendal nerve at the lateral perineum (LDI-200 probe). Parameters of frequency and duty cycle will be progressed, but power will always be set to 1%..
  Arms: Sham Low Level Laser Therapy Group

SUMMARY:
Provoked vestibulodynia (PVD) is one major subtype of vulvar pain, affecting close to one in ten women and resulting in pain during attempts at vaginal intercourse and/or attempts to insert a digit, device or tampon into the vagina. Management involves a multidisciplinary approach, through physicians, psychologists, sex therapists and physiotherapists. Low Level Laser Therapy (LLLT) is a therapeutic modality involving irradiation of injured or diseased tissue with a combination of red and infrared light. This process is thought to initiate a series of physiological reactions within the cells exposed to light at these wavelengths, leading to the restoration of normal cell structure and function. The investigators hypothesize that LLLT will be effective at reducing pain and improving sexual function among women with PVD.

The purpose of this double-blind randomized controlled trial is to assess the feasibility of using a LLLT intervention for the management of PVD in women. The aim is to determine whether there is evidence of a positive effect of LLLT, delivered using a BioFlexTM laser system (Health Canada Licence No. 7931) and a semi-standardized protocol, in terms of self-reported pain and sexual functioning, physiological responses to pressure applied at the vulvar vestibule, tonic and phasic activation of the PFM and/or corticomotor excitability to the PFMs in women with PVD with or without concurrent vaginismus (VAG) when compared to an identical treatment schedule where sham LLLT is delivered.

Women will be recruited from among eighty women with confirmed PVD and PVD+VAG who participate in a cross sectional study investigating pelvic floor muscle involvement in PVD. If they are interested in participating in this intervention study, they will be asked to consent to having their data from the cross sectional study used for the purposes of this concurrent study.

Women will be evaluated before the intervention using a battery of physical assessments and questionnaires, re-evaluated on primary outcome measures 3 weeks after initiating the intervention and then re-evaluated using the complete battery of physical assessment and questionnaires at the end of the intervention period. If we secure further funding, a medium term (12 weeks later) follow-up will be added. Physical assessment will include evaluation of pressure-pain threshold, temporal summation of pain, electromyographic (EMG) evaluation of PFM activity, responses of the PFMs to pressure applied at the vulvar vestibule using a custom electronic vulvalgesiometer, motor evoked potential threshold, amplitude, latency and the duration of cortically mediated silent period recorded from the PFMs following transcranial magnetic stimulation. The questionnaires will include the The Vulvar Pain Assessment Questionnaire (VPAQ), the Female Sexual Functioning Index, the Pain Catastrophizing Scale, the Depression Anxiety Stress Scales and the Central Sensitization Inventory. Three weeks and 12 weeks after the first start of treatment, the Global Perception of Improvement and Global patient satisfaction with treatment questionnaires will be administered. These will be repeated 12 weeks after completing treatment if funding becomes available.

DETAILED DESCRIPTION:
Vulvar pain affects the psychological and sexual health of more than one in five Canadian women, yet its pathophysiology is poorly understood. Provoked vestibulodynia (PVD) is one major subtype of vulvodynia, affecting close one in ten women and resulting in sharp, burning pain during attempts at vaginal intercourse and/or attempts to insert a digit, device or tampon into the vagina. Hypersensitivity of the vulvar vestibule is one of the key defining characteristics of PVD and, while its pathogenesis is unknown, it has been primarily attributed to inflammatory processes and hyperinnervation. Pelvic floor muscle (PFM) dysfunction has also been implicated in many forms of dyspareunia, yet the nature of this involvement also remains largely unknown.

Low Level Laser Therapy (LLLT), or photobiomodulation, is a therapeutic resource involving irradiation of injured or diseased tissue with a combination of red and infrared light. This laser is thought to initiate a series of physiological reactions within the cells exposed to light at these wavelengths, leading to the restoration of normal cell structure and function.

The purpose of this randomized controlled trial is to assess the feasibility of using a comprehensive LLLT intervention for the management of PVD in women with PVD alone (PVD) or with concurrent vaginismus (PVD+VAG). True and sham LLLT will be delivered by the BioFlexTM laser system (Health Canada License No. 7931). The aim is to determine whether there is evidence of a positive effect of LLLT delivered using a semi-standardized protocol delivered by the BioFlexTM laser in terms of primary outcomes including pain, sexual functioning and overall symptoms and secondary outcomes including changes in physiological responses to pressure applied at the vulvar vestibule, corticomotor excitability to the PFMs, and tonic activation and motor control of the PFMs.

Women will be recruited from among eighty women participating in a cross sectional study investigating pelvic floor muscle involvement in PVD. Women will therefore already have been recruited through local physiotherapists and gynecologists who have specific expertise in genital pain disorders and a diagnosis of PVD and PVD+VAG will have been confirmed through screening (Friedrich's Criteria as well as digital palpation assessment) by a gynaecologist, gynaecology resident or pelvic health physiotherapist, all with specific training on the assessment of vulvar pain. Other causes of vulvar pain, including generalized vulvodynia, infection, lichen sclerosis etc. will have been ruled out. Potential participants will be approached by the study protocol officer after they have participated in the cross sectional study and asked if they are interested in participating in this intervention study. If so, they will be asked to consent to having their data from the cross sectional study passed on to the current study.

Women will be evaluated before and after the 12-week intervention on all outcome measures, while primary outcome measures will be also evaluated after 3 weeks of intervention in both groups.

The physical assessment will be conducted by an experienced pelvic floor physiotherapist.

The evaluations will include the completion of five online questionnaires (The Vulvar Pain Assessment Questionnaire (VPAQ), Female Sexual Functioning Index, Pain Catastrophising Scale, Depression Anxiety Stress Scales, the Central Sensitization Index) and the physical assessment.

The physical assessment will involve:

1. Tampon test: participants will be provided with Original Regular Tampax Tampon and will be instructed to insert and then remove it. The participant will be instructed to report the level of pain induced through the entire insertion/removal experience on a 0-10 numeric rating scale for pain (0 meaning no pain and 10 meaning the worst pain imaginable).
2. Pressure pain threshold (PPT) will be determined involving three trials using a custom vulvalgesiometer, and will be defined as the median pressure at which women first report pain when a cotton swab tip is applied at the posterior fourchette of the vaginal introitus.
3. Temporal summation (TS) of pain: The vulvalgesiometer will again be used. A consistent pressure equivalent to the pressure that induced a pain rating of 4/10 will be applied to the posterior vaginal fourchette ten times at a rate of approximately one per second. Participants will rate their pain level on the initial and final application of this pressure using the numeric rating scale (0-10). TS will be defined as the difference in pain rating between the final and first application of the pressure.
4. Responses of the pelvic floor muscles to pressure applied at the vulvar vestibule: Women will be instrumented with electromyography (EMG) electrodes over four muscles. The superficial (bulbocavernosus and external anal sphincter) layer will be instrumented with rectangular self-adhesive gelled electrodes placed in a differential configuration on the participant's right side. The deep (pubovisceralis) PFMs will be instrumented using one custom differential suction electrode (DSE) configuration with one electrode (pole) placed on the vaginal wall overlying the muscle on the right side and the other electrode (pole) located on the anterior vaginal wall superficial to the PFMs (i.e. approx. 1.5 cm from the introitus). A common reference gelled electrode will be adhered to the skin overlying the anterior superior iliac spine on the right side. Additionally, Delsys D.E. 2.1 differential electrodes will be located over the upper trapezius muscle and over the adductor longus muscle on the right side. All EMG electrodes will be interfaced with Delsys Bagnoli-16 amplifiers (overall gain X1000, common mode rejection ratio -120dB at 60Hz; bandpass 20Hz-450Hz) and all EMG data will be sampled at 2000Hz through a 32-bit National Instruments Analog to Digital Converter (NIDAQ USB3086) and stored on a PC using Powerlab Labchart 8 Pro software. Two separate, custom vulvalgesiometers will be instrumented such that a switch that is activated when a low (25 g) or moderate (232 g) pressure is delivered. The switch (on-off) data will be recorded alongside the EMG data through the PowerLab™ software in order to separate out anticipatory activation (i.e. the EMG signal onset is before the switch is activated) from response activation (i.e. the EMG signal onset is after the switch is activated).

   The vulvalgesiometers will be used at the posterior vaginal fourchette and at the posterior aspect of the thigh. The order of the pressure application sites (vaginal fourchette vs posterior thigh) and the intensity of the pressure stimulus (low vs moderate) will be randomized using a computer generated randomization scheme. Five repetitions will be performed for each location/pressure intensity combination using a consistent inter-stimulus interval of 120 seconds. For each pressure level and site, an anticipatory response will be considered to be present on an EMG channel if, at that site, EMG activity rises two standard deviations above the noise before the pressure is applied on at least two of ten trials; while a behavioral response will be considered to be present on any EMG channel if, at that site, the EMG activity rises two standard deviations above the noise after the pressure is applied on all ten trials. For each pressure level and site, EMG response amplitudes will be recorded based on smoothed (full-wave rectified and low pass filtered using a 4th order dual-pass Butterworth filter with 3dB cut-off of 5Hz).
5. Tonic, phasic and reflex activation of the PFMs: After five minutes of rest, tonic EMG activation will be recorded from all EMG channels for a period of one minute while women are instructed to relax their PFMs as much as possible, then EMG data will be recorded throughout three trials of maximum effort PFM contractions. Next, women will be instructed on a bearing down maneuver (Valsalva) whereby they will use their diaphragm and abdominal muscles to generate an increase in intra-abdominal pressure. EMG data will be recorded from one second before the command to inhale and until 20 seconds after the command to bear down is given; three separate trials will be performed. A rest of two minutes will be given between trials and tasks to minimize the effect of fatigue, activation induced by the tasks, and/or vasovagal symptoms. Raw EMG data will be smoothed (full-wave rectified and low pass filtered using a 4th order dual-pass Butterworth filter with 3dB cut-off of 5Hz) before EMG amplitudes are determined. For tonic activation and activation during the Valsalva, mean smoothed EMG amplitude will be computed across the length over which the task is sustained. For voluntary activation, the peak smoothed EMG amplitude will be retained.
6. Corticomotor excitability of the projections to the PFMs - A Magstim® 200 system coupled with a double cone coil (96 mm loops, P/N 9902) will be used to probe the corticospinal projections to PFMs using transcranial magnetic stimulation (TMS). Participants will be fitted with a Waveguard TMS compatible cap (ANT North America Inc, WI 53719) and the vertex location will be marked at the intersection between the sagittal and coronal bisections of the head. An additional EMG channel will be added to the others already instrumented; a D.E. 2.1 electrode will be placed over the tibialis anterior muscle on the right side. With the coil at a point 2cm ventral to the vertex, magnetic stimulation intensity will be systematically increased until MEPs (50µv) are reliably evoked from the tibialis anterior muscle. The resting motor threshold (rMT) will be established using a software tool (Motor Threshold Assessment Tool 2.0) which allows fast and reliable estimation with 14 to 17 stimulations. After rMT determination, 12-20 MEPs will be recorded with participants at rest and using an intensity equivalent to 1.3 rMT. The intensity will be set at 100% maximum stimulator output in cases where the 1.3 rMT is greater than 90 % maximum stimulator output. Next the cortical silent period (cSP) will be assessed by asking participants to perform 5-10 moderate contractions of their PFMs while the TMS pulse is delivered at the same intensity (1.3 rMT) as above during the contraction. During this contraction. This will conclude the pre-intervention assessment.

After the initial assessment is complete, using concealed allocation, women will be randomized to receive either the LLLT protocol or a sham protocol, for a twelve- week intervention period using a permuted block computer-generated randomization scheme (block size 4) stratified by condition (PVD vs PVD+VAG). The participant, the protocol officer, the physiotherapists delivering the treatment and the PI will remain blinded to participant group assignment throughout the treatments and the follow-up assessment.

The intervention protocol will consist of 15 sessions provided over a 12- week period, applied by two experienced pelvic floor physiotherapists (>5 years) who have received specialized training on the application of LLLT using the Bioflex Laser system. The intervention protocol was developed in collaboration with the Clinical Director of Meditech International Rehabilitation Centers, who is also a scientific advisor to BioFlexTM Laser. Each treatment will last approximately 45 minutes and will be scheduled at the participant's convenience. During the 12- week treatment period, each participant will progress through 5 stages of treatment parameters at their own rate. The sham group will follow the same treatment steps, but the output of the laser will be at a sub-clinical intensity of 1% power. All of the steps will first include laser arrays (red and infrared light) applied to the skin overlying the sacral spine in both a horizontal and oblique placement bilaterally and the laser probe applied over the base of the spine (red and infrared light). Next, the array will be applied to the surface of the perineum (red and infrared light) followed by red light delivered by the probe at specific sites along the perineum, including the vulvar vestibule. Finally, infrared light will be applied using the probe applied to the skin overlying the branches of the pudendal nerve. Women will progress through treatment stages whereby at each stage, the same array positions and probe placement will be used but the dosage of light will be increased according to the BioFlex protocol. The laser arrays and probes will be protected with a low density polyethylene plastic cover that is compliant with the Food and Drug Administration (FDA) and United States Department of Health and Human Services (USDA) regulations. Each cover will be discarded after a single use. A mindfulness-based meditation will be provided during each assessment through noise cancelling headphones interfaced to a PC playing an audio CD. To ensure that the physiotherapists delivering the treatment remain blinded to the treatment being delivered, the real and sham (A and B) protocols have been entered into the Bioflex Laser system by the supplier and verified by a physiotherapist who is not involved in the study to ensure that they are correct. In this way none of the investigators will know which protocol (A or B) is the real treatment, and black towels will be used to cover the arrays while the treatment is delivered such that any differences in light intensity will not be visible.

Three weeks after initiating the intervention, women will repeat the five on-line questionnaires, the tampon test, PPT testing, TS testing as well as Global Perception of Improvement and Global satisfaction with treatment questionnaires, reporting to a research assistant who will remain blinded to treatment assignment. After the final treatment session (12 weeks), women will repeat these on-line questionnaires as well as the tampon test, PPT testing, TS testing, tonic and voluntary activation, anticipatory and behavioural responses, and the TMS protocol, administered by the same, blinded physiotherapist who performed the initial assessment.

After all follow-up visits are complete, women, and the research assistants, will learn whether they received the real or sham LLLT therapy, and those who received sham therapy will be invited to begin the real intervention. If follow-on funding becomes available, all women will be re-evaluated at 12 weeks following the initial therapy on all outcomes.

All outcomes will first be tested for normality using the Shapiro-Wilks test. If all outcomes are normally distributed, they will be compared between the using repeated measures (RM) ANOVA models. The Global perception of improvement will be compared between group (intervention vs control) and time (3 weeks after beginning the intervention, 12 weeks after beginning the intervention, 12 weeks after completing the intervention if available) using a three-way RM ANOVA and including condition (PVD, PVD+VAG) as a nested effect. The other outcomes will be compared between groups using three-way RM ANOVAs including group (intervention, control) and time (pre-intervention, post-intervention, 12 weeks later if available) as main effects, and including condition (PVD, PVD+VAG) as a nested effect. Alpha=0.05 will be used for all tests and effect sizes will be computed based on group means and standard deviations. Adherence rates will be recorded and intent to treat analyses are planned for participants who drop out or are lost to follow-up. For outcomes that are not normally distributed, equivalent non-parametric tests will be used wherever possible.

The sample size is based on the only pilot study that tested the therapeutic effect of LLLT on women with PVD, this study reported a significant, positive effect on pain reported during attempts at sexual intercourse among women with PVD (n=18) treated using LLLT when compared to controls (n=16) who received sham LLLT. They found that participants who received the treatment were more likely than controls to report significant or complete improvement in their pain (p=0.042) on verbal report at follow-up, a scale similar to the "Global Perception of Improvement" scale as described in this proposal. Using this result, a post-hoc power analysis (Minitab, V. 18) suggested that a sample size of 16 per group will be adequate to see a significant difference in treatment outcomes between women who receive the LLLT intervention and those who receive the sham intervention. The results of the pilot study did not demonstrate a significant treatment effect in any of their objective parameters. For example, post-hoc power analysis (MinitabTM v. 18) estimates that 154 participants per group would be required to detect a difference between treatment and control using the tampon test as the primary outcome. Given that the LLLT intervention proposed here is far more comprehensive than that used in the only pilot study published so far, there may be a greater effect associated with the proposed protocol as compared to the effect seen in the published pilot study.

ELIGIBILITY:
Inclusion Criteria

* Biologically born female older than eighteen years
* Premenopausal
* Not currently pregnant or pregnancy in the past six months
* No metal or electronic implants near neck or head
* No neurological condition such as stroke, multiple sclerosis, spinal cord injury, epilepsy or history of epilepsy in the family
* No tendency to faint
* Signs and symptoms consistent with provoked vestibulodynia alone or provoked vestibulodynia plus vaginismus

Exclusion Criteria

* gynaecologist cannot insert a single digit intravaginally and thus the participant would be unlikely able to tolerate the assessment procedures
* other evidence of conditions that may cause vulvar pain such as active lichen sclerosis, fissures, or infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Global perception of improvement | 3 weeks (during intervention)
  The Global perception of improvement is a single question through which participants provide a ordinal rating based on their overall perception of improvement attributed to the intervention.
  Much Better, Better, About the same, Worse, Much worse.
  Higher ratings is associated with better outcomes.
Global perception of improvement | 12 weeks (following intervention)
  The Global perception of improvement is a single question through which participants provide a ordinal rating based on their overall perception of improvement attributed to the intervention.
  Much Better, Better, About the same, Worse, Much worse.
  Higher ratings is associated with better outcomes.
Global perception of improvement | 12 weeks after intervention (if funding becomes available)
  The Global perception of improvement is a single question through which participants provide a ordinal rating based on their overall perception of improvement attributed to the intervention.
  Much Better, Better, About the same, Worse, Much worse.
  Higher ratings is associated with better outcomes.
The Vulvar Pain Assessment Questionnaire (VPAQ)Inventory:COMPREHENSIVE (FULL) VERSION | Baseline
  Designed to assess: pain quality, the temporal nature of the pain, associated symptoms, pain intensity, emotional/cognitive functioning, physical functioning, coping strategies, and interpersonal functioning.
  Core Domains: Consists of 63 items:8 questions assessing the onset, location, temporal pattern, degree of burning pain, and associated symptoms of vulvar pain, along with six subscales. Subscales are composed of 55 items rated on 5-point scales with anchors tailored to the nature of the questions being asked:
  1. Pain severity
  2. Emotional response
  3. Cognitive response
  4. Life interference
  5. Sexual function interference
  6. Self-stimulation/penetration interference
  Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms
The Vulvar Pain Assessment Questionnaire (VPAQ)Inventory:COMPREHENSIVE (FULL) VERSION | 3 weeks (during intervention)
  Designed to assess: pain quality, the temporal nature of the pain, associated symptoms, pain intensity, emotional/cognitive functioning, physical functioning, coping strategies, and interpersonal functioning.
  Core Domains: Consists of 63 items:8 questions assessing the onset, location, temporal pattern, degree of burning pain, and associated symptoms of vulvar pain, along with six subscales. Subscales are composed of 55 items rated on 5-point scales with anchors tailored to the nature of the questions being asked:
  1. Pain severity
  2. Emotional response
  3. Cognitive response
  4. Life interference
  5. Sexual function interference
  6. Self-stimulation/penetration interference
  Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms
The Vulvar Pain Assessment Questionnaire (VPAQ)Inventory:COMPREHENSIVE (FULL) VERSION | 12 weeks (following intervention)
  Designed to assess: pain quality, the temporal nature of the pain, associated symptoms, pain intensity, emotional/cognitive functioning, physical functioning, coping strategies, and interpersonal functioning.
  Core Domains: Consists of 63 items:8 questions assessing the onset, location, temporal pattern, degree of burning pain, and associated symptoms of vulvar pain, along with six subscales. Subscales are composed of 55 items rated on 5-point scales with anchors tailored to the nature of the questions being asked:
  1. Pain severity
  2. Emotional response
  3. Cognitive response
  4. Life interference
  5. Sexual function interference
  6. Self-stimulation/penetration interference
  Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms
The Vulvar Pain Assessment Questionnaire (VPAQ) Inventory:COMPREHENSIVE (FULL) VERSION | 12 weeks after intervention (if funding becomes available)
  Designed to assess: pain quality, the temporal nature of the pain, associated symptoms, pain intensity, emotional/cognitive functioning, physical functioning, coping strategies, and interpersonal functioning.
  Core Domains: Consists of 63 items:8 questions assessing the onset, location, temporal pattern, degree of burning pain, and associated symptoms of vulvar pain, along with six subscales. Subscales are composed of 55 items rated on 5-point scales with anchors tailored to the nature of the questions being asked:
  1. Pain severity
  2. Emotional response
  3. Cognitive response
  4. Life interference
  5. Sexual function interference
  6. Self-stimulation/penetration interference
  Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms
Pain rating during the tampon test | Baseline
  The participants will be provided with Original Regular Tampax Tampon and will be instructed to insert and then remove it. After, they will be asked to record the degree of pain during the entire insertion/removal experience in a 11-point numerical rating scale (NRS) with anchors of 0 (no pain at all) to 10 (worst pain imaginable).
Pain rating during the tampon test | 3 weeks (during the intervention)
  The participants will be provided with Original Regular Tampax Tampon and will be instructed to insert and then remove it. After, they will be asked to record the degree of pain during the entire insertion/removal experience in a 11-point numerical rating scale (NRS) with anchors of 0 (no pain at all) to 10 (worst pain imaginable).
Pain rating during the tampon test | 12 weeks (immediately after the intervention)
  The participants will be provided with Original Regular Tampax Tampon and will be instructed to insert and then remove it. After, they will be asked to record the degree of pain during the entire insertion/removal experience in a 11-point numerical rating scale (NRS) with anchors of 0 (no pain at all) to 10 (worst pain imaginable).
Pain rating during the tampon test | 12 weeks later (if funding becomes available)
  The participants will be provided with Original Regular Tampax Tampon and will be instructed to insert and then remove it. After, they will be asked to record the degree of pain during the entire insertion/removal experience in a 11-point numerical rating scale (NRS) with anchors of 0 (no pain at all) to 10 (worst pain imaginable)..
Pressure pain threshold (PPT) at the posterior vaginal fourchette | Baseline
  PPT will be determined using a custom vulvalgesiometer and will be defined as the average pressure at which women first report pain when the cotton swab tip is applied at 6 o' clock position of the vaginal introitus. The vulvalgesiometer will also be used to evaluate TS of pain when the pressure measured before will be applied ten times at a rate of approximately one per second at the same location on the vestibule. Participants will rate their pain level on the initial and final application of this pressure using the same numeric rating scale (0-10).
Pressure pain threshold (PPT) at the posterior vaginal fourchette | 3 weeks (during the intervention)
  PPT will be determined using a custom vulvalgesiometer and will be defined as the average pressure at which women first report pain when the cotton swab tip is applied at 6 o' clock position of the vaginal introitus. The vulvalgesiometer will also be used to evaluate TS of pain when the pressure measured before will be applied ten times at a rate of approximately one per second at the same location on the vestibule. Participants will rate their pain level on the initial and final application of this pressure using the same numeric rating scale (0-10).
Pressure pain threshold (PPT) at the posterior vaginal fourchette | 12 weeks (following intervention)
  PPT will be determined using a custom vulvalgesiometer and will be defined as the average pressure at which women first report pain when the cotton swab tip is applied at 6 o' clock position of the vaginal introitus. The vulvalgesiometer will also be used to evaluate TS of pain when the pressure measured before will be applied ten times at a rate of approximately one per second at the same location on the vestibule. Participants will rate their pain level on the initial and final application of this pressure using the same numeric rating scale (0-10).
Pressure pain threshold (PPT) at the posterior vaginal fourchette | 12 weeks after intervention (if funding becomes available)
  PPT will be determined using a custom vulvalgesiometer and will be defined as the average pressure at which women first report pain when the cotton swab tip is applied at 6 o' clock position of the vaginal introitus. The vulvalgesiometer will also be used to evaluate TS of pain when the pressure measured before will be applied ten times at a rate of approximately one per second at the same location on the vestibule. Participants will rate their pain level on the initial and final application of this pressure using the same numeric rating scale (0-10).
Temporal summation of pain | Baseline
  Difference between pain reported on first application of pressure at the vulvar vestibule, delivered through a vulvalgesiometer, and the pain reported after the tenth application of that same pressure
Temporal summation of pain | 3 weeks (during the intervention)
  Difference between pain reported on first application of pressure at the vulvar vestibule, delivered through a vulvalgesiometer, and the pain reported after the tenth application of that same pressure
Temporal summation of pain | 12 weeks (after the intervention)
  Difference between pain reported on first application of pressure at the vulvar vestibule, delivered through a vulvalgesiometer, and the pain reported after the tenth application of that same pressure
Temporal summation of pain | 12 weeks later (if funding becomes available)
  Difference between pain reported on first application of pressure at the vulvar vestibule, delivered through a vulvalgesiometer, and the pain reported after the tenth application of that same pressure

SECONDARY OUTCOMES:
Global Patient satisfaction with treatment | 3 weeks (during intervention)
  Global patient satisfaction with treatment is a single question through which participants provide a ordinal rating based on their satisfaction with the intervention.
  Completely, Somewhat, Not at all.
  Higher ratings is associated with better outcomes.
Global Patient satisfaction with treatment | 12 weeks (following intervention)
  Global patient satisfaction with treatment is a single question through which participants provide a ordinal rating based on their satisfaction with the intervention.
  Completely, Somewhat, Not at all.
  Higher ratings is associated with better outcomes.
Global Patient satisfaction with treatment | 12 weeks after intervention (if funding becomes available)
  Global patient satisfaction with treatment is a single question through which participants provide a ordinal rating based on their satisfaction with the intervention.
  Completely, Somewhat, Not at all.
  Higher ratings is associated with better outcomes.
Female Sexual Function Index (FSFI) | Baseline
  This is a 19-item validated questionnaire for assessing the key dimension of sexual function in women, considered a gold standard for evaluation of sexual function. It assesses six domains: desire, arousal , lubrification, orgasm, satisfaction, and pain. All scores are totaled for a maximum of 36. Higher scores represents better sexual function. A score ≤26.55 has been set as a cutoff to identify those at risk for sexual dysfunction.
Female Sexual Function Index (FSFI) | 12 weeks (following intervention)
  This is a 19-item validated questionnaire for assessing the key dimension of sexual function in women, considered a gold standard for evaluation of sexual function. It assesses six domains: desire, arousal , lubrification, orgasm, satisfaction, and pain. All scores are totaled for a maximum of 36. Higher scores represents better sexual function. A score ≤26.55 has been set as a cutoff to identify those at risk for sexual dysfunction.
Female Sexual Function Index (FSFI) | 12 weeks after intervention (if funding becomes available)
  This is a 19-item validated questionnaire for assessing the key dimension of sexual function in women, considered a gold standard for evaluation of sexual function. It assesses six domains: desire, arousal , lubrification, orgasm, satisfaction, and pain. All scores are totaled for a maximum of 36. Higher scores represents better sexual function. A score ≤26.55 has been set as a cutoff to identify those at risk for sexual dysfunction.
Motor evoked potential (MEP) peak to peak amplitude (µV) | Baseline
  Transcranial magnetic stimulation outcome will be determined for all participants and compared among groups. A Magstim® 200 system coupled with a double coil (96 mm loops, P/N 9902) will be used to probe the corticospinal projections to PFMs. MEPs will be ensemble averaged to generate estimates of MEP peak to peak amplitude (µV).
Motor evoked potential (MEP) peak to peak amplitude (µV) | 12 weeks (immediately after the intervention)
  Transcranial magnetic stimulation outcome will be determined for all participants and compared among groups. A Magstim® 200 system coupled with a double coil (96 mm loops, P/N 9902) will be used to probe the corticospinal projections to PFMs. MEPs will be ensemble averaged to generate estimates of MEP peak to peak amplitude (µV).
Motor evoked potential (MEP) peak to peak amplitude (µV) | 12 weeks later (if funding becomes available)
  Transcranial magnetic stimulation outcome will be determined for all participants and compared among groups. A Magstim® 200 system coupled with a double coil (96 mm loops, P/N 9902) will be used to probe the corticospinal projections to PFMs. MEPs will be ensemble averaged to generate estimates of MEP peak to peak amplitude (µV).
Cortical silent period (ms) | Baseline
  Transcranial magnetic stimulation outcome will be determined for all participants and compared among groups. A Magstim® 200 system coupled with a double coil (96 mm loops, P/N 9902) will be used to probe the corticospinal projections to PFMs. MEP cortical silent period (cSP) will be measured from individual trials and then averaged.
Cortical silent period (ms) | 12 weeks (immediately after the intervention)
  Transcranial magnetic stimulation outcome will be determined for all participants and compared among groups. A Magstim® 200 system coupled with a double coil (96 mm loops, P/N 9902) will be used to probe the corticospinal projections to PFMs. MEP cortical silent period (cSP) will be measured from individual trials and then averaged.
Cortical silent period (ms) | 12 weeks later (if funding becomes available)
  Transcranial magnetic stimulation outcome will be determined for all participants and compared among groups. A Magstim® 200 system coupled with a double coil (96 mm loops, P/N 9902) will be used to probe the corticospinal projections to PFMs. MEP cortical silent period (cSP) will be measured from individual trials and then averaged.
Pain Catastrophizing Scale | Baseline
  This is a reliable and valid scale to measure of catastrophizing. The scores from this questionnaire is predictors of intensity of physical and emotional distress. It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
Pain Catastrophizing Scale | 12 weeks (after the intervention)
  This is a reliable and valid scale to measure of catastrophizing. The scores from this questionnaire is predictors of intensity of physical and emotional distress. It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
Pain Catastrophizing Scale | 12 weeks later (if funding becomes available)
  This is a reliable and valid scale to measure of catastrophizing. The scores from this questionnaire is predictors of intensity of physical and emotional distress. It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
Depression Anxiety Stress Scale (DASS) | Baseline
  This is a 42-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress. Each one contains 14 items, divided into subscales of 2-5 items with similar content. The DASS have been shown to have high internal consistency and to yield meaningful discriminations in a variety of settings.
  A higher score on the DASS indicates greater severity or frequency of these negative emotional symptoms. The maximum score is 126.
Depression Anxiety Stress Scale (DASS) | 3 weeks (during the intervention)
  This is a 42-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress. Each one contains 14 items, divided into subscales of 2-5 items with similar content. The DASS have been shown to have high internal consistency and to yield meaningful discriminations in a variety of settings.
  A higher score on the DASS indicates greater severity or frequency of these negative emotional symptoms. The maximum score is 126.
Depression Anxiety Stress Scale (DASS) | 12 weeks (after the intervention)
  This is a 42-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress. Each one contains 14 items, divided into subscales of 2-5 items with similar content. The DASS have been shown to have high internal consistency and to yield meaningful discriminations in a variety of settings.
  A higher score on the DASS indicates greater severity or frequency of these negative emotional symptoms. The maximum score is 126.
Depression Anxiety Stress Scale (DASS) | 12 weeks later (if funding becomes available)
  This is a 42-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress. Each one contains 14 items, divided into subscales of 2-5 items with similar content. The DASS have been shown to have high internal consistency and to yield meaningful discriminations in a variety of settings.
  A higher score on the DASS indicates greater severity or frequency of these negative emotional symptoms. The maximum score is 126.
Central sensitization index | Baseline
  The Central Sensitisation Inventory (CSI) is a self-report outcome measure designed to identify patients who have symptoms that may be related to central sensitisation (CS) or central sensitivity syndromes (CSS). Part A includes 25 questions related to common CSS symptoms.
  Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression. CSI severity levels have been established for part A: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100.
Central sensitization index | 12 weeks (after the intervention)
  The Central Sensitisation Inventory (CSI) is a self-report outcome measure designed to identify patients who have symptoms that may be related to central sensitisation (CS) or central sensitivity syndromes (CSS). Part A includes 25 questions related to common CSS symptoms.
  Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression. CSI severity levels have been established for part A: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100.
Central sensitization index | 12 weeks later (if funding becomes available)
  The Central Sensitisation Inventory (CSI) is a self-report outcome measure designed to identify patients who have symptoms that may be related to central sensitisation (CS) or central sensitivity syndromes (CSS). Part A includes 25 questions related to common CSS symptoms.
  Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression. CSI severity levels have been established for part A: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100.
The Vulvar Pain Assessment Questionnaire - Supplemental Domains | Baseline
  Supplemental Domains Pain Descriptors (VPAQdesc). This pain descriptor scale contains the most common words used to describe chronic vulvar pain.
  1. Burning/stinging pain
  2. Incisive pain
  3. Sensitivity
  Coping Strategies (VPAQcope). This scale addresses some common coping strategies that are utilized by women with vulvar pain.
  1. Distraction/relaxation strategies
  2. Problem-solving strategies
  Partner Factors (VPAQpartner). This 24-item scale encompasses how romantic partners/spouses may be impacted by/respond to vulvar pain experienced by one partner.
  1. Negative response
  2. Support seeking
  3. Impact on relationship
  4. Sexual communication
  Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms
The Vulvar Pain Assessment Questionnaire - Supplemental Domains | 3 weeks (during intervention)
  Supplemental Domains Pain Descriptors (VPAQdesc). This pain descriptor scale contains the most common words used to describe chronic vulvar pain.
  1. Burning/stinging pain
  2. Incisive pain
  3. Sensitivity
  Coping Strategies (VPAQcope). This scale addresses some common coping strategies that are utilized by women with vulvar pain.
  1. Distraction/relaxation strategies
  2. Problem-solving strategies
  Partner Factors (VPAQpartner). This 24-item scale encompasses how romantic partners/spouses may be impacted by/respond to vulvar pain experienced by one partner.
  1. Negative response
  2. Support seeking
  3. Impact on relationship
  4. Sexual communication Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms
The Vulvar Pain Assessment Questionnaire - Supplemental Domains | 12 weeks (following intervention)
  Supplemental Domains Pain Descriptors (VPAQdesc). This pain descriptor scale contains the most common words used to describe chronic vulvar pain.
  1. Burning/stinging pain
  2. Incisive pain
  3. Sensitivity
  Coping Strategies (VPAQcope). This scale addresses some common coping strategies that are utilized by women with vulvar pain.
  1. Distraction/relaxation strategies
  2. Problem-solving strategies
  Partner Factors (VPAQpartner). This 24-item scale encompasses how romantic partners/spouses may be impacted by/respond to vulvar pain experienced by one partner.
  1. Negative response
  2. Support seeking
  3. Impact on relationship
  4. Sexual communication
  Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms
The Vulvar Pain Assessment Questionnaire - Supplemental Domains | 12 weeks after intervention (if funding becomes available)
  Supplemental Domains Pain Descriptors (VPAQdesc). This pain descriptor scale contains the most common words used to describe chronic vulvar pain.
  1. Burning/stinging pain
  2. Incisive pain
  3. Sensitivity
  Coping Strategies (VPAQcope). This scale addresses some common coping strategies that are utilized by women with vulvar pain.
  1. Distraction/relaxation strategies
  2. Problem-solving strategies
  Partner Factors (VPAQpartner). This 24-item scale encompasses how romantic partners/spouses may be impacted by/respond to vulvar pain experienced by one partner.
  1. Negative response
  2. Support seeking
  3. Impact on relationship
  4. Sexual communication
  Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms

OTHER OUTCOMES:
Tonic activation of the pelvic floor muscles (PFMs) | Baseline
  Mean smoothed, rectified activation amplitude of the PFMs recorded through electromyography while the muscles remain at rest.
Tonic activation of the pelvic floor muscles (PFMs) | 12 weeks (after intervention)
  Mean smoothed, rectified activation amplitude of the PFMs recorded through electromyography while the muscles remain at rest.
Tonic activation of the pelvic floor muscles (PFMs) | 12 weeks later (if funding becomes available)
  Mean smoothed, rectified activation amplitude of the PFMs recorded through electromyography while the muscles remain at rest.
Maximum voluntary activation of the pelvic floor muscles (PFMs) | Baseline
  Mean smoothed, rectified activation amplitude of the PFMs recorded through electromyography while participants attempt a maximum voluntary activation of their PFMs
Maximum voluntary activation of the pelvic floor muscles (PFMs) | 12 weeks (after intervention)
  Mean smoothed, rectified activation amplitude of the PFMs recorded through electromyography while participants attempt a maximum voluntary activation of their PFMs
Maximum voluntary activation of the pelvic floor muscles (PFMs) | 12 weeks later (if funding becomes available)
  Mean smoothed, rectified activation amplitude of the PFMs recorded through electromyography while participants attempt a maximum voluntary activation of their PFMs
Activation of the pelvic floor muscles (PFMs) during a bearing down maneuver | Baseline
  Mean smoothed, rectified activation amplitude of the PFMs recorded through electromyography while participants perform a bearing down maneuver
Activation of the pelvic floor muscles (PFMs) during a bearing down maneuver | 12 weeks (after intervention)
  Mean smoothed, rectified activation amplitude of the PFMs recorded through electromyography while participants perform a bearing down maneuver
Activation of the pelvic floor muscles (PFMs) during a bearing down maneuver | 12 weeks later (if funding becomes available)
  Mean smoothed, rectified activation amplitude of the PFMs recorded through electromyography while participants perform a bearing down maneuver
Anticipatory responses (ms) to pressure applied at the vulvar vestibule | Baseline
  The proportion of women in each group who demonstrate anticipatory responses of the PFMs to impeding pressure applied at the vulvar vestibule will be determined for each group. Participants will be deemed to have anticipatory responses if electromyiographic signals recorded from the PFMs precede the application of pressure. A vulvagesiometer will be employed using a response-dependent methodology. The vulvagesiometer will be used to apply low (25g) and moderate (232g) pressure to the posterior vaginal fourchette or to the posterior thigh.
Anticipatory responses (ms) to pressure applied at the vulvar vestibule | 12 weeks (after the intervention)
  The proportion of women in each group who demonstrate anticipatory responses of the PFMs to impeding pressure applied at the vulvar vestibule will be determined for each group. Participants will be deemed to have anticipatory responses if electromyiographic signals recorded from the PFMs precede the application of pressure. A vulvagesiometer will be employed using a response-dependent methodology. The vulvagesiometer will be used to apply low (25g) and moderate (232g) pressure to the posterior vaginal fourchette or to the posterior thigh.
Anticipatory responses (ms) to pressure applied at the vulvar vestibule | 12 weeks later (if funding becomes available)
  The proportion of women in each group who demonstrate anticipatory responses of the PFMs to impeding pressure applied at the vulvar vestibule will be determined for each group. Participants will be deemed to have anticipatory responses if electromyiographic signals recorded from the PFMs precede the application of pressure. A vulvagesiometer will be employed using a response-dependent methodology. The vulvagesiometer will be used to apply low (25g) and moderate (232g) pressure to the posterior vaginal fourchette or to the posterior thigh.
Behavioural responses (µV) to pressure applied at the vulvar vestibule | Baseline
  The proportion of women in each group who demonstrate behavioural responses of the PFMs to pressure applied at the vulvar vestibule will be determined for each group. Participants will be deemed to have behavioural responses if the activation of the PFMs (or other muscles) occurs after the pressure is applied. A vulvagesiometer will be employed using a response-dependent methodology. The vulvagesiometer will be used to apply low (25g) and moderate (232g) pressure to the posterior vaginal fourchette or to the posterior thigh.
Behavioural responses (µV) to pressure applied at the vulvar vestibule | 12 weeks (after the intervention)
  The proportion of women in each group who demonstrate behavioural responses of the PFMs to pressure applied at the vulvar vestibule will be determined for each group. Participants will be deemed to have behavioural responses if the activation of the PFMs (or other muscles) occurs after the pressure is applied. A vulvagesiometer will be employed using a response-dependent methodology. The vulvagesiometer will be used to apply low (25g) and moderate (232g) pressure to the posterior vaginal fourchette or to the posterior thigh.
Behavioural responses (µV) to pressure applied at the vulvar vestibule | 12 weeks later (if funding becomes available)
  The proportion of women in each group who demonstrate behavioural responses of the PFMs to pressure applied at the vulvar vestibule will be determined for each group. Participants will be deemed to have behavioural responses if the activation of the PFMs (or other muscles) occurs after the pressure is applied. A vulvagesiometer will be employed using a response-dependent methodology. The vulvagesiometer will be used to apply low (25g) and moderate (232g) pressure to the posterior vaginal fourchette or to the posterior thigh.
Adherence to the intervention protocol | 12 weeks (after the intervention)
  Attendance of laser treatment visits will be tracked.

CONTACTS AND LOCATIONS:
Overall Officials: Linda McLean, Principal Investigator — University of Ottawa
Locations (1):
- McLean Function Measurement Lab, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Spreadsheets will be provided by email upon request and based on the planned use of the data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 10 years after the publication of the study results.
Access Criteria: Planned use of data for systematic review or meta-analysis.

REFERENCES:
- [Background] Harlow BL, Stewart EG. A population-based assessment of chronic unexplained vulvar pain: have we underestimated the prevalence of vulvodynia? J Am Med Womens Assoc (1972). 2003 Spring;58(2):82-8. PMID 12744420
- [Background] Spoelstra SK, Dijkstra JR, van Driel MF, Weijmar Schultz WC. Long-term results of an individualized, multifaceted, and multidisciplinary therapeutic approach to provoked vestibulodynia. J Sex Med. 2011 Feb;8(2):489-96. doi: 10.1111/j.1743-6109.2010.01941.x. PMID 20646179
- [Background] Vallinga MS, Spoelstra SK, Hemel IL, van de Wiel HB, Weijmar Schultz WC. Transcutaneous electrical nerve stimulation as an additional treatment for women suffering from therapy-resistant provoked vestibulodynia: a feasibility study. J Sex Med. 2015 Jan;12(1):228-37. doi: 10.1111/jsm.12740. Epub 2014 Nov 12. PMID 25388372
- [Background] Goldstein AT, Pukall CF, Brown C, Bergeron S, Stein A, Kellogg-Spadt S. Vulvodynia: Assessment and Treatment. J Sex Med. 2016 Apr;13(4):572-90. doi: 10.1016/j.jsxm.2016.01.020. Epub 2016 Mar 25. PMID 27045258
- [Background] Migliario M, Sabbatini M, Mortellaro C, Reno F. Near infrared low-level laser therapy and cell proliferation: The emerging role of redox sensitive signal transduction pathways. J Biophotonics. 2018 Nov;11(11):e201800025. doi: 10.1002/jbio.201800025. Epub 2018 Aug 16. PMID 29722183
- [Background] Passarella S. He-Ne laser irradiation of isolated mitochondria. J Photochem Photobiol B. 1989 Aug;3(4):642-3. doi: 10.1016/1011-1344(89)80090-9. No abstract available. PMID 2507765
- [Background] Ailioaie C, Lupusoru-Ailioaie LM. Beneficial effects of laser therapy in the early stages of rheumatoid arthritis onset. Laser Ther 11(2):79-87, 1999.
- [Background] Foster DC, Beth Kotok M, Huang LS, Watts A, Oakes D, Howard FM, Stodgell CJ, Dworkin RH. The tampon test for vulvodynia treatment outcomes research: reliability, construct validity, and responsiveness. Obstet Gynecol. 2009 Apr;113(4):825-832. doi: 10.1097/AOG.0b013e31819bda7c. PMID 19305326
- [Background] Pukall CF, Young RA, Roberts MJ, Sutton KS, Smith KB. The vulvalgesiometer as a device to measure genital pressure-pain threshold. Physiol Meas. 2007 Dec;28(12):1543-50. doi: 10.1088/0967-3334/28/12/008. Epub 2007 Dec 3. PMID 18057518
- [Background] McLean L, Brooks K. What Does Electromyography Tell Us About Dyspareunia? Sex Med Rev. 2017 Jul;5(3):282-294. doi: 10.1016/j.sxmr.2017.02.001. Epub 2017 Mar 18. PMID 28330675
- [Background] Brostrom S. Motor evoked potentials from the pelvic floor. Neurourol Urodyn. 2003;22(7):620-37. doi: 10.1002/nau.10151. PMID 14595605
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Meyer-Bahlburg HF, Dolezal C. The female sexual function index: a methodological critique and suggestions for improvement. J Sex Marital Ther. 2007 May-Jun;33(3):217-24. doi: 10.1080/00926230701267852. PMID 17454519
- [Background] Sullivan MJL, et al. The Pain Catastrophizing Scale: Development and validation. Psychological Assessment 7, 524-532, 1995.
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Antony, Martin & Bieling, Peter & Cox, Brian & Enns, Murray & Swinson, Richard. (1998). Psychometric properties of the 42-item and 21-item versions of the Depression Anxiety Stress Scales in clinical groups and a community sample. Psychological Assessment. 10. 176-181. 10.1037/1040-3590.10.2.176.
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Burgio KL, Goode PS, Richter HE, Locher JL, Roth DL. Global ratings of patient satisfaction and perceptions of improvement with treatment for urinary incontinence: validation of three global patient ratings. Neurourol Urodyn. 2006;25(5):411-7. doi: 10.1002/nau.20243. PMID 16652380
- [Background] Pukall, C.F., Cahill, C.M. New Developments in the Pathophysiology of Genital Pain: Role of Central Sensitization. Curr Sex Health Rep 6, 11-19 (2014) doi:10.1007/s11930-013-0007-1.
- [Background] Reissing ED, Brown C, Lord MJ, Binik YM, Khalife S. Pelvic floor muscle functioning in women with vulvar vestibulitis syndrome. J Psychosom Obstet Gynaecol. 2005 Jun;26(2):107-13. doi: 10.1080/01443610400023106. PMID 16050536
- [Background] Gentilcore-Saulnier E, McLean L, Goldfinger C, Pukall CF, Chamberlain S. Pelvic floor muscle assessment outcomes in women with and without provoked vestibulodynia and the impact of a physical therapy program. J Sex Med. 2010 Feb;7(2 Pt 2):1003-22. doi: 10.1111/j.1743-6109.2009.01642.x. Epub 2010 Jan 6. PMID 20059663
- [Background] Morin M, et al. Dynamometric assessment of the pelvic floor muscle function in women with and without provoked vestibulodynia. Int Urogynecol J 2010: 21: S336-S37
- [Background] Morin M, Bergeron S, Khalife S, Mayrand MH, Binik YM. Morphometry of the pelvic floor muscles in women with and without provoked vestibulodynia using 4D ultrasound. J Sex Med. 2014 Mar;11(3):776-85. doi: 10.1111/jsm.12367. Epub 2013 Nov 6. PMID 24344835
- [Background] McLean L, Thibault-Gagnon S, Brooks K, Goldfinger C, Pukall C, Chamberlain S. Differences in Pelvic Morphology Between Women With and Without Provoked Vestibulodynia. J Sex Med. 2016 Jun;13(6):963-71. doi: 10.1016/j.jsxm.2016.04.066. PMID 27215690
- [Background] Dargie EE, Chamberlain SM, Pukall CF. Provoked Vestibulodynia: Diagnosis, Self-Reported Pain, and Presentation During Gynaecological Examinations. J Obstet Gynaecol Can. 2017 Mar;39(3):145-151. doi: 10.1016/j.jogc.2017.01.001. PMID 28343555
- [Background] Lev-Sagie A, Kopitman A, Brzezinski A. Low-Level Laser Therapy for the Treatment of Provoked Vestibulodynia-A Randomized, Placebo-Controlled Pilot Trial. J Sex Med. 2017 Nov;14(11):1403-1411. doi: 10.1016/j.jsxm.2017.09.004. Epub 2017 Sep 29. PMID 28970071
- [Derived] I Antonio F, Pukall C, McLean L. Photobiomodulation therapy for the treatment of vulvar pain among those with provoked vestibulodynia: a randomized controlled trial. J Sex Med. 2025 Apr 15;22(4):579-587. doi: 10.1093/jsxmed/qdaf011. PMID 39940084